CLINICAL TRIAL: NCT00873249
Title: Effect of Daily SMS Reminders on Medication Adherence to Oral Antipsychotics in Patients With Schizophrenia
Brief Title: Effect of Daily Short Message System (SMS) Reminders on Medication Adherence to Oral Antipsychotics in Patients With Schizophrenia
Acronym: SMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Diez, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2007/3
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Therapeutic adherence; Short message system; Mobile phone
MeSH Terms: conditions — Schizophrenia; Treatment Adherence and Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a 6-month, multicenter, randomized study to assess the effect of daily SMS reminders sent during 3 months in the adherence to oral antipsychotic treatment in stabilized outpatients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years
* With a diagnosis of schizophrenia (DSM-IV TR criteria)
* Stabilized out-patients
* Under oral antipsychotic monotherapy

Exclusion Criteria:

* Administration of a depot antipsychotic drug
* Suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stabilized outpatients with a diagnosis of schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Morisky Green Questionnaire | baseline, at months 3 and 6

SECONDARY OUTCOMES:
Clinical Global Impression- Schizophrenia (CGI-SCH) | baseline, at months 3 and 6
Register of Adherence to Treatment (RAT) | baseline, at months 3 and 6

CONTACTS AND LOCATIONS:
Locations (25):
- Spain (25):
  - Research Site, Alicante, Alicante
  - Research Site, Almería, Almeria
  - Research Site, Barcelona, Barcelona
  - Research Site, Berga, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Burgos, Burgos
  - Research Site, Santander, Cantabria
  - Research Site, Córdoba, Cordoba
  - Research Site, Granada, Granada
  - Research Site, León, Leon
  - Research Site, Lleida, Lerida
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Murcia, Murcia
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Oviedo
  - Research Site, Palma Mallorca, Palma Mallorca
  - Research Site, Salamanca, Salamanca
  - Research Site, Seville, Sevilla
  - Research Site, Tarragona, Tarragona
  - Research Site, Toledo, Toledo
  - Research Site, Valencia, Valencia
  - Research Site, Valladolid, Valladolid
  - Research Site, Zamora, Zamora
  - Research Site, Calatayud, Zaragoza